CLINICAL TRIAL: NCT01321541
Title: A Randomized Multicenter Study Comparing Pixantrone + Rituximab With Gemcitabine + Rituximab in Patients With Aggressive B-cell Non-Hodgkin Lymphoma Who Have Relapsed After Therapy With CHOP-R or an Equivalent Regimen and Are Ineligible for Stem Cell Transplant
Brief Title: Comparison of Pixantrone + Rituximab With Gemcitabine + Rituximab in Patients With Aggressive B-cell Non-Hodgkin Lymphoma or Follicular Grade 3 Lymphoma Who Have Relapsed After Therapy and Are Not Eligible for Stem Cell Transplant
Acronym: PIX-R
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIX306 (PIX-R Trial)
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-09

CONDITIONS: Diffuse Large B-cell Lymphoma; de Novo DLBCL; DLBCL Transformed From Indolent Lymphoma; Follicular Grade 3 Lymphoma
Keywords: non-hodgkin lymphoma; DLBCL; relapsed; aggressive NHL; Diffuse large B-cell lymphoma; Rituximab; Rituxan; Pixantrone; NHL; non hodgkin's lymphoma; de novo DLBCL; DLBCL transformed from Indolent Lymphoma; Follicular Grade 3 Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Recurrence | interventions — pixantrone; Rituximab; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pixantrone + Rituximab (Experimental): Pixantrone and Rituximab
  Interventions: Drug: Pixantrone + Rituximab
- Gemcitabine + Rituximab (Active Comparator): Gemcitabine and Rituximab
  Interventions: Drug: Gemcitabine + Rituximab

INTERVENTIONS:
Drug: Pixantrone + Rituximab — Pixantrone + Rituximab: Rituximab 375 mg/m2 IV on day 1 and pixantrone 50 mg/m2 (equivalent to 85mg/m2 pixantrone dimaleate)IV on days 1, 8, and 15. Regimen is given in 28-day cycles. Up to 6 cycles may be administered.
  Arms: Pixantrone + Rituximab
Drug: Gemcitabine + Rituximab — Gemcitabine + Rituximab: Rituximab 375 mg/m2 IV on day 1 and gemcitabine 1000 mg/m2 IV on days 1, 8, and 15. Regimen is given in 28-day cycles. Up to 6 cycles may be administered.
  Arms: Gemcitabine + Rituximab

SUMMARY:
The purpose of this study is to evaluate the efficacy of Pixantrone + Rituximab compared to Gemcitabine + Rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL), or follicular grade 3 lymphoma.

DETAILED DESCRIPTION:
Eligible patients will be randomized to treatment with pixantrone plus rituximab or gemcitabine plus rituximab in up to six 28-day cycles. At the time patients experience progressive disease during study treatment, early follow- up, or intermediate follow-up, they enter the survival follow up period. Patients who complete study treatment or discontinue study treatment for any other reason will participate in the follow-up periods.

Early Follow-Up: After treatment completion or discontinuation, patient will enter a 24-week follow-up period.

Intermediate Follow-Up: After completing the 24-week early follow-up period, patient will enter an additional 72-week follow-up period.

Survival Follow-Up: All patients will be monitored for survival.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DLBCL (de novo DLBCL, or transformed from indolent lymphoma) or follicular grade 3 lymphoma on the basis of tissue biopsy.
2. Patients with de novo DLBCL must have received 1-3 treatment regimens for DLBCL. Patients with follicular grade 3 lymphoma must have received 1-3 treatment regimens for follicular lymphoma (any grade). Patients with DLBCL transformed from indolent lymphoma must have received at least 1-4 treatment regimens for NHL.
3. Received rituximab containing a multi-agent therapy for the treatment of NHL.
4. Not eligible for high-dose chemotherapy and stem cell transplant.
5. Patients with DLBCL transformed from indolent lymphoma must have had a complete or partial response to a therapy for NHL lasting at least 12 weeks.

Exclusion Criteria:

1. Primary refractory de novo DLBCL or primary refractory follicular grade 3 lymphoma, defined as documented progression within 12 weeks of the last cycle of the first-line multi-agent regimen.
2. Prior treatment with cumulative dose of doxorubicin or equivalent exceeding 450 mg/m2
3. Any experimental therapy ≤ 28 days prior to randomization
4. Other malignancy within last 5 years except for the following: curatively treated basal cell/squamous cell skin cancer, carcinoma in situ of the cervix, superficial transitional cell bladder carcinoma, or in situ ductal carcinoma of the breast after complete resection
5. Any contraindication or known allergy or hypersensitivity to any study drugs
6. Concomitant therapy with any anticancer agents, immunosuppressive agents, other investigational anticancer therapies. Low-dose corticosteroids for the treatment of non cancer-related illnesses are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2011-04-20 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simran B Singh, MS, GWCP, Study Director — Sr. Director, Clinical Operations
Locations (127):
- United States (47):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Highlands Oncology Group, Bentonville, Arkansas
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - George Washington University Department of Medicine, Washington D.C., District of Columbia
  - Integrated Community Oncology Network-St. Vincent's, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside, Jacksonville, Florida
  - Integrated Community Oncology Network, Orange Park, Florida
  - Carle Physician Group, Danville, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Foundation Physician Services, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Baptist Hospital East, Louisville, Kentucky
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, PC, Bethesda, Maryland
  - Cancer & Hematology Center of Western Michigan, Grand Rapids, Michigan
  - Metro Minnesota CCOP-Unity Hospital, Fridley, Minnesota
  - Metro Minnesota CCOP-St. Johns, Maplewood, Minnesota
  - Metro Minnesota Community Clinical Oncology Program, Saint Louis Park, Minnesota
  - Metro Minnesota CCOP-Regions Hospital, Saint Paul, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Hematology-Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - North Shore Hematology/Oncology Associates, East Setauket, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Gabrail Cancer Center, Dover, Ohio
  - Toledo Clinical Cancer Center, Toledo, Ohio
  - Mercy Cancer Center at St. Anne's, Toledo, Ohio
  - Toledo Clinic Cancer Center-Toledo, Toledo, Ohio
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Upstate Oncology Associates, Greenville, South Carolina
  - South Carolina Cancer Specialists, Hardeeville, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Cancer Care Centers of South Texas-HOAST, New Braunfels, Texas
  - Cancer Care Centers of South Texas-HOAST, San Antonio, Texas
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - Saint Vincent Hospital Green Bay Oncology, Green Bay, Wisconsin
  - Green Bay Oncology-St. Mary's Hospital MC, Green Bay, Wisconsin
- Austria (3):
  - Medical University Innsbruck, Department of Internal Medicine V (Hematology and Oncology), Innsbruck
  - Hospital Elisabethinen Linz, Internal Department 1 - Hemato-Oncology, Linz
  - Hanusch Hospital, Department of Internal Medicine III, Vienna
- Belgium (3):
  - Saint Luc University Hospital, Department of Hematology, Brussels
  - General Hospital Delta, Hematology Department, Roeselare
  - General Hospital Turnhout, Hematology Department, Turnhout
- Bulgaria (6):
  - UMHAT "Sveti Georgi", Plovdiv, Clinical Hematology Clinic, Plovdiv
  - UMHAT "Sveti Georgi", Plovdiv, Department of Medical Oncology, Plovdiv
  - MHAT "Tokuda Hospital Sofia", Hematology Clinic, Sofia
  - University Multiprofile Hospital for Active Treatment "Sveti Ivan Rilski", Department of Clinical Hematology, Sofia
  - Specialized Hospital For Active Treatment Of Hematological Diseases, Sofia, Clinical Hematology Clinic, Sofia
  - MHAT Hristo Botev, Vratsa, First Department of Internal Medicine, Vratsa
- Czechia (5):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Hradec Kralove, 4th Department of Internal Medicne, Clinical Hematology, Hradec Králové
  - University Hospital Ostrava, Institute of Clinical Hematology, Ostrava
  - University Hospital Kralovske Vinohrady, Department of Clinical Hematology, Prague
  - General University Hospital in Prague, 1st Department of Internal Medicine - Department of Hematology, Prague
- Aalborg University Hospital, Department of Hematology, Aalborg, Denmark
- France (8):
  - Service d'hématologie clinique, Avenue Laennec Salouel, Amiens
  - Centre hopitalier de la cote basque, Bayonne
  - Centre hospitalier de Beziers, Béziers
  - Polyclinique de Bordeaux nord Acquitaine, Bordeaux
  - Centre hospitalier du Mans, Le Mans
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Saint Quentin Hospital Center, Department of Oncology-Hematology, Saint-Quentin
  - Hautepierre Hospital, Department of Hematology and Oncology, Strasbourg
- Germany (8):
  - Gemeinschaftspraxis Drs. Klausmann, Aschaffenburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinik Köln, Cologne
  - Klinik für Innere Medizin III, Frankfurt (a.M.)
  - Universitaetsklinikum Halle, Halle
  - St. Marien Hospital Hamm, Hamm
  - Klinikum Nürnberg Nord, Nuremberg
  - Klinikum Mutterhaus der Borromäerinnen, Trier
- Hungary (3):
  - St. Istvan and St. Laszlo Hospital of Budapest, Budapest
  - University of Debrecen, Debrecen
  - Moritz Kaposi General Hospital, Kaposvár
- Italy (9):
  - University Hospital "Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi", Ancona
  - Bologna University Hospital Authority St. Orsola-Malpighi Polyclinic, Bologna
  - Scientific Institute of Romagna for the Study and Treatment of Cancer (I.R.S.T.) S.R.L., Meldola
  - "Ospedali Riuniti Villa Sofia-Cervello" Hospital, Palermo
  - Romagna Local Health Authority (AUSL Romagna) - "Santa Maria delle Croci", Ravenna
  - Romagna Local Health Authority (AUSL Romagna) - "Infermi" Hospital, Rimini
  - Siena University Hospital Authority Santa Maria alle Scotte Polyclinic, Siena
  - Santa Maria Hospital, Terni
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
- Poland (8):
  - Independent Public Healthcare Facility Municipal Hospital Group, Chorzów
  - Marine Hospital of Polish Red Cross, Department of Chemotheraphy, Gdynia
  - Silesia Medical University, Department of Hematology and Bone Marrow Transplantation, Katowice
  - Malopolskie Medical Center S.C. , Department of Hematology, Krakow
  - Nicolaus Copernicus Memorial Provincial Specialist Hospital in Lodz, Lodz
  - Oncology Center of Lublin Land, Department of Clinical Oncology, Lublin
  - Institute of Hematology and Transfusion Medicine, Clinic of Hematology, Warsaw
  - Wroclaw Medical University, Department and Clinic of Hematology, Blood Neoplasms and Bone Marrow Transplantation, Wroclaw
- Romania (3):
  - Rapid Diagnosis Polyclinic SA, Brasov
  - Fundeni Clinical Institute Center for Hematology and Bone Marrow Transplantation, Bucharest
  - Bucharest University Emergency Hospital, Hematology Clinic, Bucharest
- Russia (6):
  - Federal State Public Institution: Main Military Clinical Hospital n.a. N.N. Burdenko of the Russian Ministry of Defense, Moscow
  - Moscow State Budget Medical Institution: City Clinical Hospital n.a. S.P.Botkin, Moscow
  - State Medical Institution: Republican Hospital named after V.A. Baranov, Petrozavodsk
  - St. Petersburg Clinical Research and Practical Center for Specialized Types of Medical Care, Saint Petersburg
  - State Healthcare Institution: Republican Clinical Oncology Center, Ufa
  - State Budget Healthcare Institution of Sverdlovsk region: Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Slovakia (4):
  - University Hospital with Outpatient Clinic F.D. Roosevelt Banska Bystrica, Department of Hematology, Banská Bystrica
  - National Cancer Institute, Department of Hematology and Transfusiology, Bratislava
  - University Hospital Martin, Department of Hematology and Transfusiology, Martin
  - J. A. Reiman University Hospital with Polyclinic in Presov, Prešov
- Spain (6):
  - A Coruña University Hospital, A Coruña
  - Hospital Universitario Vall Hebrón, Barcelona
  - Hospital Iniversitario Puerta del Mar, Cadiz
  - Institut Català de Oncologia (ICO), Hospital Dr Trueta, Girona
  - Hospital Iniversitario La Paz, Madrid
  - Hospital Universitario Araba, Vitoria-Gasteiz
- Ukraine (4):
  - Cherkasy Regional Oncology Center, Regional Treatment and Diagnostic Hematology Center, Cherkasy
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - National Institute of Cancer, Kyiv
  - State Institution: Institute of Blood Pathology and Transfusion Medicine, Lviv
- United Kingdom (3):
  - Beatson West of Scotland Cancer Center, Glasgow
  - St. George's Healthcare NHS Trust, London
  - Christie Hospital, Department of Medical Oncology, Manchester

REFERENCES:
- [Result] Pettengell R, Dlugosz-Danecka M, Andorsky D, Belada D, Georgiev P, Quick D, Singer JW, Singh SB, Pallis A, Egorov A, Salles G. Pixantrone plus rituximab versus gemcitabine plus rituximab in patients with relapsed aggressive B-cell non-Hodgkin lymphoma not eligible for stem cell transplantation: a phase 3, randomized, multicentre trial (PIX306). Br J Haematol. 2020 Jan;188(2):240-248. doi: 10.1111/bjh.16255. Epub 2019 Dec 27. PMID 31879945
- [Derived] Belada D, Georgiev P, Dakhil S, Inhorn LF, Andorsky D, Beck JT, Quick D, Pettengell R, Daly R, Dean JP, Pavlyuk M, Failloux N, Hubel K. Pixantrone-rituximab versus gemcitabine-rituximab in relapsed/refractory aggressive non-Hodgkin lymphoma. Future Oncol. 2016 Aug;12(15):1759-68. doi: 10.2217/fon-2016-0137. Epub 2016 Apr 20. PMID 27093976

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
Started | 155 | 157
Completed | 72 | 61
Not Completed | 83 | 96

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab | Total
Number analyzed (Participants) | 155 | 157 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 30 | 66
  >=65 years | 119 | 127 | 246
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 90 | 176
  Male | 69 | 67 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 147 | 155 | 302
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
IPI Score [Count of Participants; unit: Participants] — International Prognostic Index (IPI) Score Calculation:
  IPI Points Characteristic:
  1pt - Age > 60 years
  1pt - Performance Status 2, 3 or 4
  1pt - NHL Stage III or IV
  1pt - Elevated LDH
  1pt - More than 1 extranodal site
  Maximum Score Possible: 5
  IPI Score 0-2 = better outcome IPI Score 3 or greater = worse outcome
  Participants
    IPI Score 0-2 | 73 | 73 | 146
    IPI Score 3 or more | 82 | 84 | 166
Ann Arbor Stage [Count of Participants; unit: Participants] — Ann Arbor Staging System I = Involvement of a single lymph node or a single extranodal organ/site, II = Involvement of ≥ 2 lymph node regions on the same side of the diaphragm, or localized involvement of an extranodal site/organ, III = Involvement of lymph node regions on both sides of the diaphragm, which may be also accompanied by local involvement of an extranodal organ/site, IV = Diffuse or disseminated involvement of one or more distant extranodal organs with or without associated lymph node involvement I-III = better outcome, IV = worse outcome
  Participants
    I-III | 81 | 76 | 157
    IV | 74 | 81 | 155
Number ofprior lines of therapy [Count of Participants; unit: Participants]
  0-2 | 137 | 139 | 276
  3 or more | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time of randomization to the date of disease progression or death due to any cause (whichever occurs first)
Time Frame: From the date of randomization to the date of progressive disease or death due to any cause (whichever is first reported) (Up to 100 weeks)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
Number analyzed (Participants) | 155 | 157
Months | 7.3 [5.2 to 8.4] | 6.3 [4.4 to 8.1]

2. Secondary Outcome: Overall Survival
Description: Overall survival is from randomization to death due to any cause
Time Frame: From date of randomization to the date of the patient's death due to any cause (Up to 100 weeks)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
Number analyzed (Participants) | 155 | 157
Months | 13.3 [10.1 to 19.8] | 19.6 [12.4 to 31.9]

3. Secondary Outcome: Complete Response Rate
Description: CRR is defined as the proportion of patients who achieve a Complete Response (CR) without additional therapy. CR is defined as the disappearance of all target lesions.
Time Frame: From date of randomization to the date of the patient's death due to any cause (Up to 100 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
Number analyzed (Participants) | 155 | 157
Participants | 55 | 34

4. Secondary Outcome: Overall Response Rate
Description: ORR is defined as the proportion of patients who achieve a CR or PR without additional therapy.
Time Frame: From date of randomization to the date of the patient's death due to any cause (Up to 100 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
Number analyzed (Participants) | 155 | 157
percentage of patients | 61.9 [53.8 to 69.6] | 43.9 [36.0 to 52.1]

5. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAE) Related to Study Drug
Description: The number of Participants with Treatment Emergent Adverse Events (TEAE) related to study drug (pixantrone or gemcitabine)
Time Frame: From date of randomization to the date of the patient's death due to any cause (Up to 100 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
Number analyzed (Participants) | 153 | 146
Participants | 140 | 140

6. Other Pre Specified Outcome: Individual Concentration-time Profiles of Patients Will be Compared to Existing Data Using Simulations (Visual Predictive Checks)
Description: To characterize the PK profile of pixantrone when co-administered with rituximab. Plasma samples for PK analysis will be collected relative to the D-1 dose of pixantrone in one of the 6 treatment cycles for each participating patient. The goal is to enroll approx. 20 patients, active at 20 sites- Beatson West of Scotland Cancer Center, Uni. Hospital Kralovske Vinohrady, Uni. Hospital Hradec Kralove Hematooncology, Hospital Nuernberg, St. Marien Hospital Hamm, Puerta del Mar Hospital, Tokuda Hospital Sofia, National Center of Hematology & Transfusiology, UMHAT "SV. IVAN RILSKI", Moritz Kaposi General Hospital, Uni. of Debrecen, Polish Red Cross Marine Hospital, Kharkiv Regional Clinical Oncology Center, National Inst. of Cancer Ukraine, Cherkasy Regional Oncology Center, Inst. of Blood Pathology & Transfusion Medicine, Uni. Hospital Martin, National Onclogy Inst., Uni. Hospital with Outpatient Clinic F.D. Roosevelt Banska Bystrica, Uni. Hospital J.A. Reiman Presov
Time Frame: within 1 hour of initiation of infusion to 24-48 hours after start of pixantrone infusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: To Generate Individual Secondary PK Parameters (eg, Exposure, Half-life Etc.) Using Descriptive Statistics
Description: as for outcome 6
Time Frame: within 1 hour of initiation of infusion to 24-48 hours after start of pixantrone infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent until 30 days after the last dose of study treatment. (Up to 100 weeks)
Description: Safety will be assessed by monitoring and recording adverse events, serious adverse events, cardiac, hematologic and blood chemistry parameters, vital signs, performance status, and any abnormal findings observed on physical examinations
Arm/Group | Pixantrone + Rituximab | Gemcitabine + Rituximab
All-Cause Mortality (participants affected / at risk) | 12/153 | 16/149
Serious Adverse Events (participants affected / at risk) | 59/153 | 57/149
Other Adverse Events (participants affected / at risk) | 153/153 | 148/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pixantrone + Rituximab (N=153) | Gemcitabine + Rituximab (N=149)
Pneumonia (Infections and infestations) | 8 (8) | 4 (4)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal bacteremia (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Cytotoxic cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 8 (8)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Disseminated large cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pixantrone + Rituximab (N=153) | Gemcitabine + Rituximab (N=149)
Neutropenia (Blood and lymphatic system disorders) | 105 (105) | 87 (87)
Anaemia (Blood and lymphatic system disorders) | 37 (37) | 67 (67)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (23) | 95 (95)
Leukopenia (Blood and lymphatic system disorders) | 12 (12) | 19 (19)
Lymphopenia (Blood and lymphatic system disorders) | 10 (10) | 5 (5)
Fatigue (General disorders) | 45 (45) | 34 (34)
Pyrexia (General disorders) | 20 (20) | 30 (30)
Asthenia (General disorders) | 20 (20) | 18 (18)
Oedema peripheral (General disorders) | 19 (19) | 30 (30)
Chills (General disorders) | 11 (11) | 10 (10)
Nausea (Gastrointestinal disorders) | 38 (38) | 22 (22)
Constipation (Gastrointestinal disorders) | 35 (35) | 20 (20)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 19 (19)
Vomiting (Gastrointestinal disorders) | 21 (21) | 17 (17)
Stomatitis (Gastrointestinal disorders) | 16 (16) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (29) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 15 (15) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 10 (10)
Pneumonia (Infections and infestations) | 10 (10) | 9 (9)
Urinary tract infection (Infections and infestations) | 9 (9) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 28 (28) | 16 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (14) | 11 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (10) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 19 (19)
Dizziness (Nervous system disorders) | 15 (15) | 7 (7)
Headache (Nervous system disorders) | 12 (12) | 6 (6)
Dysgeusia (Nervous system disorders) | 11 (11) | 3 (3)
Weight decreased (Investigations) | 12 (12) | 4 (4)
Ejection fraction decreased (Investigations) | 8 (8) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 10 (10)
Platelet count decreased (Investigations) | 1 (1) | 9 (9)
Alanine aminotransferase increased (Investigations) | 0 (0) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7)
Hypotension (Musculoskeletal and connective tissue disorders) | 17 (17) | 6 (6)
Hypertension (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (10)
Anxiety (Psychiatric disorders) | 8 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01321541/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT01321541/SAP_001.pdf